CLINICAL TRIAL: NCT04950816
Title: Examining the Feasibility and Acceptability of a Tailored Version of a Mindfulness-Based Intervention (MBI) Among Youth Experiencing Homelessness (YEH) Aged 18-25 Years Old
Brief Title: Examining the Feasibility and Acceptability of a Tailored Version of a Mindfulness-Based Intervention (MBI) Among Youth Experiencing Homelessness (YEH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Diane Santa Maria, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSC-SN-20-0466 (Aim 3 Pilot); 5R34AT010672-03 (NIH)
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stress, Emotional
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tailored MBI (.b) (Experimental)
  Interventions: Behavioral: tailored MBI (.b)
- attention control condition (Active Comparator)
  Interventions: Behavioral: attention control condition

INTERVENTIONS:
Behavioral: tailored MBI (.b) — The session will include brief didactic presentations, videos, and mindfulness practice followed by inquiry. We anticipate that sessions will take place twice a week. Sessions will be held on site at the Covenant House Texas (CHT) shelter in a quiet, designated learning space to ease access to sessions for the participants and to assure access to shelter staff (e.g., social workers and case managers) and services (e.g., food and shelter). CHT has onsite, weekday clinical and mental health care and established protocols for accessing needed resources 24/7. Selection criteria for the interventionist include maintaining a personal mindfulness practice for at least two years, trained in .b, and prior experience working with high-risk youth. The interventionist will receive additional training in Trauma-Informed Care as well as study procedures.
  Arms: tailored MBI (.b)
Behavioral: attention control condition — Participants will receive no training in MBI or meditation. Topics covered may include physical activity, nutrition, managing weight, understanding adolescence, personal care, avoiding tobacco, alcohol, and drugs though this will be finalized in YR-1 with the HYWG and advisory panel. The HT program will be led by a positive adult instructor with training in health education or a related field and experience working with YEH.
  Arms: attention control condition

SUMMARY:
The purpose of this study is to conduct a trial of the tailored Mindfulness- Based Intervention (MBI) (.b) vs. attention control to test real-world feasibility and acceptability of this tailored Mindfulness - Based Intervention (MBI) in youth experiencing homelessness (YEH).

ELIGIBILITY:
Inclusion Criteria:

* homeless youth receiving services at one of the recruitment sites in Houston, Texas area at the time of enrollment
* English speaking
* able to participate for the entire study period (i.e., not moving during the study)

Exclusion Criteria:

* overtly exhibiting symptoms of severe, untreated mental illness criteria
* not staying at the shelter
* currently experiencing homelessness or unstable housing

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane M Santa Maria, DrPH,MSN,RN,PHNA-BC,FSAHM,FAAN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 121 participants were screened. Of those, 90 met the inclusion criteria and were enrolled.
Period: Overall Study
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Started | 45 | 45
Completed Immediately After Intervention (About 2 to 4 Weeks After Baseline) | 36 | 39
Completed 3 Month Post Intervention Follow up | 31 | 28
Completed 6 Month Post Intervention Follow up | 25 | 24
Completed | 25 | 24
Not Completed | 20 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tailored MBI (.b) | Attention Control Condition | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.05 (1.86) | 21.90 (1.81) | 21.48 (1.88)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 10 | 17 | 27
  Male | 29 | 27 | 56
  Transgender Female | 2 | 0 | 2
  Transgender Male | 2 | 0 | 2
  Non-binary/ non-conforming | 1 | 1 | 2
  Other (unspecified) | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 13 | 26
  Not Hispanic or Latino | 32 | 32 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 19 | 28 | 47
  White | 12 | 4 | 16
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Emotion Regulation as Measured by Difficulties in Emotion Regulation Scale (DERS)
Description: The DERS is a 36-item questionnaire, and each item is scored from 1(almost never)-5 (almost always). The 36 items were added to generate a scale from 36 to 180, a higher score indicates greater problem with emotion regulation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 45 | 45
score on a scale | 93.18 (26.41) | 82.62 (23.42)

2. Primary Outcome: Emotion Regulation as Measured by Difficulties in Emotion Regulation Scale (DERS)
Description: as for outcome 1
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: Data were not collected from 4 participants in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 86.03 (21.82) | 94.74 (21.19)

3. Primary Outcome: Emotion Regulation as Measured by Difficulties in Emotion Regulation Scale (DERS)
Description: as for outcome 1
Time Frame: 3 months post intervention
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey. Data were not collected from 1 participant in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
score on a scale | 85.4 (22.25) | 91.56 (19.64)

4. Primary Outcome: Emotion Regulation as Measured by Difficulties in Emotion Regulation Scale (DERS)
Description: as for outcome 1
Time Frame: 6 months post intervention
Population: Data were not collected from 1 participant in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 23
score on a scale | 90.36 (24.21) | 94.26 (17.17)

5. Primary Outcome: Mindfulness as Measured by Child and Adolescent Mindfulness Measure (CAMM)
Description: The CAMM is a 10 item questionnaire and each item is scored from 0(never true)-4 (always true). The 10 items were added to generate a scale from 0 to 40, a higher score indicates higher levels of mindfulness
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 45 | 45
score on a scale | 23.84 (9.3) | 27.38 (11.26)

6. Primary Outcome: Mindfulness as Measured by Child and Adolescent Mindfulness Measure (CAMM)
Description: as for outcome 5
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 26.89 (9.47) | 24.31 (10.41)

7. Primary Outcome: Mindfulness as Measured by Child and Adolescent Mindfulness Measure (CAMM)
Description: as for outcome 5
Time Frame: 3 months post intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
score on a scale | 28.73 (9.08) | 27.74 (10.61)

8. Primary Outcome: Mindfulness as Measured by Child and Adolescent Mindfulness Measure (CAMM)
Description: as for outcome 5
Time Frame: 6 months post intervention
Population: Data were not collected from 2 participants in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 22
score on a scale | 25.92 (9.2) | 30.36 (9.39)

9. Primary Outcome: Mindfulness as Measured by Cognitive and Affective Mindfulness Scale-Revised (CAMS-R)
Description: The CAMS-R is a 12-item measure and each item is scored from 1( rarely/not at all)-4(almost always). Higher values reflect greater mindful qualities
Time Frame: Baseline, immediately after intervention (about 2 to 4 weeks after baseline),3 months post intervention,6 months post intervention
Population: Data were not collected for this outcome measure because the Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) was not administered to participants. Instead, the Child and Adolescent Mindfulness Measure (CAMM) was used to assess Mindfulness. As a result, no participants received the CAMS-R, and no data were collected for this outcome measure. Therefore, zero participants were analyzed for this outcome. Data from the CAMM are reported under a different outcome measure.
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Self-Compassion as Measured by Self-Compassion Scale (SCS)
Description: The Self-Compassion Scale (SCS) total score ranges from 1 to 5, higher score indicating greater self compassion..
Time Frame: Baseline
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 44 | 45
score on a scale | 3.06 (0.47) | 3.21 (0.44)

11. Primary Outcome: Self-Compassion as Measured by Self-Compassion Scale (SCS)
Description: The Self-Compassion Scale (SCS) total score ranges from 1 to 5, higher score indicating greater self compassion.
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey. Data were not collected from 4 participants in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 35 | 35
score on a scale | 3.11 (0.60) | 3.05 (0.33)

12. Primary Outcome: Self-Compassion as Measured by Self-Compassion Scale (SCS)
Description: The Self-Compassion Scale (SCS) total score ranges from 1 to 5, higher score indicating greater self compassion.
Time Frame: 3 months post intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
score on a scale | 3.20 (0.60) | 3.15 (0.37)

13. Primary Outcome: Self-Compassion as Measured by Self-Compassion Scale (SCS)
Description: The Self-Compassion Scale (SCS) total score ranges from 1 to 5, higher score indicating greater self compassion.
Time Frame: 6 months post intervention
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 22
score on a scale | 3.23 (0.43) | 3.06 (0.25)

14. Primary Outcome: Stress as Measured by Perceived Stress Scale (PSS)
Description: The PSS is a 10 item questionnaire and each item is scored from 0(never)-4(very often). The 10 items were added to generate a scale from 0 to 40, higher score indicating a higher perceived stress.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 44 | 45
score on a scale | 20.59 (5.51) | 18.31 (7.15)

15. Primary Outcome: Stress as Measured by Perceived Stress Scale (PSS)
Description: as for outcome 14
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 18.64 (6.2) | 17.97 (5.4)

16. Primary Outcome: Stress as Measured by Perceived Stress Scale (PSS)
Description: as for outcome 14
Time Frame: 3 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 31 | 28
score on a scale | 16.58 (4.97) | 18.07 (4.65)

17. Primary Outcome: Stress as Measured by Perceived Stress Scale (PSS)
Description: as for outcome 14
Time Frame: 6 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 23
score on a scale | 18.48 (4.64) | 18.65 (2.92)

18. Primary Outcome: Feasibility as Assessed by the Percentage of Participants Enrolled in the Study
Description: Percentage of participants who met study eligibility criteria who enroll (provide informed consent) in the study
Time Frame: Baseline
Population: This outcome measure includes only participants who were enrolled in the pilot trial.
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Screened: All subjects who were screened
Arm/Group | All Subjects Screened
Number analyzed (Participants) | 121
Participants | 90

19. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Adhere to Treatment
Description: Number of participants who adhere to treatment is measured by the number of participants who attended at least 3 of 5 group sessions.
Time Frame: 6 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 45 | 45
Participants | 35 | 41

20. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Completed the 3 Months Follow up
Time Frame: 3 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 45 | 45
Participants | 31 | 28

21. Primary Outcome: Feasibility as Assessed by the Number of Participants Who Completed the 6 Months Follow up
Time Frame: 6 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 45 | 45
Participants | 25 | 24

22. Primary Outcome: Acceptability as Assessed by the Credibility and Expectancy Questionnaire - Expectancy Subscale
Description: The Credibility and Expectancy Questionnaire (CEQ) was used to assess the acceptability of the intervention. All participants completed both subscales: the credibility subscale and the expectancy subscale. Each subscale total score ranges from 0 to 10, with higher scores indicating greater perceived acceptability. The expectancy subscale is reported.
Time Frame: 6 months post intervention
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 32 | 29
score on a scale | 7.05 (2.28) | 6.09 (2.74)

23. Secondary Outcome: Social Connectedness as Measured Social Connectedness Scale
Description: The scale is a 8 item questionnaire and each item is scored from 1(strongly disagree)-6(strongly agree). The 8 items were added to generate a scale from, 8 to 48, a higher score indicating more connectedness to others.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 44 | 45
score on a scale | 30.36 (11.24) | 31.20 (12.54)

24. Secondary Outcome: Social Connectedness as Measured Social Connectedness Scale
Description: as for outcome 23
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 27.64 (11.79) | 30.46 (11.07)

25. Secondary Outcome: Social Connectedness as Measured Social Connectedness Scale
Description: as for outcome 23
Time Frame: 3 months post intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
score on a scale | 30.4 (12.13) | 31.59 (12.56)

26. Secondary Outcome: Social Connectedness as Measured Social Connectedness Scale
Description: as for outcome 23
Time Frame: 6 months post intervention
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 22
score on a scale | 26.32 (10.69) | 32.26 (12.03)

27. Secondary Outcome: Depression as Measured by Short Mood and Feelings Questionnaire (SMFQ)
Description: The scale is a 13 item questionnaire and each item is scored from 0(not true)-2(true),higher score indicating worse outcome
Time Frame: Baseline, immediately after intervention (1day after baseline),3 months post intervention,6 months post intervention
Population: Data were not collected for this outcome measure because the Short Mood and Feelings Questionnaire (SMFQ) was not administered to participants. Instead, the Patient Health Questionnaire-9 (PHQ-9) was used to assess Depression. As a result, no participants received the SMFQ, and no data were collected for this outcome measure. Therefore, zero participants were analyzed for this outcome. Data from the PHQ-9 are reported under a different outcome measure.
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Anxiety as Measured by Spielberger State-Trait Anxiety Inventory
Description: This scale is a 40 item questionnaire, each question is scored from 1(very much so)-4 (not at all), a higher score indicates a worse outcome
Time Frame: Baseline, immediately after intervention (1day after baseline),3 months post intervention,6 months post intervention
Population: Data were not collected for this outcome measure because the Spielberger State-Trait Anxiety Inventory was not administered to participants. Instead, the Generalized Anxiety Disorder (GAD) Scale was used to assess Anxiety. As a result, no participants received the Spielberger State-Trait Anxiety Inventory and no data were collected for this outcome measure. Therefore, zero participants were analyzed for this outcome. Data from the GAD Scale are reported under a different outcome measure.
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Vulnerability as Measured by Psychological Vulnerability Scale
Description: The Psychological Vulnerability Scale is a 6 item questionnaire. Each item is scored from 1 (does not describe me at all) to 5 (describes me very well). The 6 items were added to generate a scale from 6 to 30, a higher score indicates more vulnerability.
Time Frame: Baseline
Population: Data were not collected from 2 participants in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 43 | 45
score on a scale | 14.81 (5.1) | 13.16 (6.35)

30. Secondary Outcome: Vulnerability as Measured by Psychological Vulnerability Scale
Description: as for outcome 29
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 13.92 (5.84) | 15.34 (5.79)

31. Secondary Outcome: Vulnerability as Measured by Psychological Vulnerability Scale
Description: as for outcome 29
Time Frame: 3 months post intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
score on a scale | 12.57 (4.85) | 12.85 (6.67)

32. Secondary Outcome: Vulnerability as Measured by Psychological Vulnerability Scale
Description: as for outcome 29
Time Frame: 6 months post intervention
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 22
score on a scale | 14.2 (6.96) | 12.27 (6.33)

33. Secondary Outcome: Risk Seeking as Measured by Balloon Analogue Risk Task (BART)
Description: The Balloon Analogue Risk Task (BART) is a computerized measure of risk taking behavior. Each click causes the balloon to incrementally inflate and money to be added to a counter up until some threshold, at which point the balloon is over inflated and explodes. The primary score used to measure BART performance is the adjusted average number of pumps on unexploded balloons, with higher scores indicative of greater risk-taking propensity
Time Frame: Baseline, immediately after intervention (about 2-4 weeks after baseline),3 months post intervention,6 months post intervention
Population: Data were not collected for this outcome measure because the Balloon Analogue Risk Task (BART) was not administered to participants. Instead, the Risk Propensity Scale was used to assess Risk Seeking. As a result, no participants received the Balloon Analogue Risk Task (BART), and no data were collected for this outcome measure. Therefore, zero participants were analyzed for this outcome. Data from the Risk Propensity Scale are reported under a different outcome measure.
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Distress as Measured by Kessler Psychological Distress Scale (K10)
Description: This is a 10-item questionnaire,each item is scored from 1(none of the time)-5(all of the time) for a total score ranging from 10-50 and a higher score indicating worse outcome
Time Frame: Baseline, immediately after intervention (1day after baseline),3 months post intervention,6 months post intervention
Population: Data were not collected for this outcome measure because the Kessler Psychological Distress Scale (K10) was not administered to participants. Instead, the PROMIS Item Bank v.1.0-Emotional Distress was used to assess Distress. As a result, no participants received the K10 , and no data were collected for this outcome measure. Therefore, zero participants were analyzed for this outcome. Data from the PROMIS Item Bank v.1.0-Emotional Distress are reported under a different outcome measure.
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Number of Participants Who Are Sexually Active
Description: A single item question was used to assess this outcome. The item asked whether or not you ever had sexual intercourse. The number of participants who answered yes is reported.
Time Frame: Baseline
Population: Data were not collected from 3 participants in the tailored MBI (.b) arm because they did not complete the survey. Data were not collected from 2 participants in the attention control condition arm because they did not complete the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 42 | 43
Participants | 30 | 24

36. Secondary Outcome: Number of Participants Who Are Sexually Active
Description: as for outcome 35
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: Data were not collected from 5 participants in the attention control condition arm because they did not complete the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 34
Participants | 28 | 21

37. Secondary Outcome: Number of Participants Who Are Sexually Active
Description: as for outcome 35
Time Frame: 3 months post intervention
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the question. Data were not collected from 1 participant in the attention control condition arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
Participants | 18 | 18

38. Secondary Outcome: Number of Participants Who Are Sexually Active
Description: as for outcome 35
Time Frame: 6 months post intervention
Population: Data were not collected from 3 participants in the attention control condition arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 21
Participants | 20 | 16

39. Secondary Outcome: Number of Participants Who Ever Used Drugs or Substances (Marijuana, Prescription Pain Medicine Without a Prescription, Synethic Marijuana, Cocaine, Inhalants, Heroin, Meth, Ecstasy, Injection Drugs)
Description: A single item question was used to assess this outcome. The item listed various drug substances and asked whether any of those listed had been used in their life. The number of participants who answered yes is reported.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 45 | 45
Participants | 35 | 34

40. Secondary Outcome: Number of Participants Who Ever Used Drugs or Substances (Marijuana, Prescription Pain Medicine Without a Prescription, Synethic Marijuana, Cocaine, Inhalants, Heroin, Meth, Ecstasy, Injection Drugs)
Description: as for outcome 39
Time Frame: Immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 36
Participants | 29 | 28

41. Secondary Outcome: Number of Participants Who Ever Used Drugs or Substances (Marijuana, Prescription Pain Medicine Without a Prescription, Synethic Marijuana, Cocaine, Inhalants, Heroin, Meth, Ecstasy, Injection Drugs)
Description: as for outcome 39
Time Frame: 3 months post intervention
Population: as for outcome 37
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
Participants | 22 | 20

42. Secondary Outcome: Number of Participants Who Ever Used Drugs or Substances (Marijuana, Prescription Pain Medicine Without a Prescription, Synethic Marijuana, Cocaine, Inhalants, Heroin, Meth, Ecstasy, Injection Drugs)
Description: as for outcome 39
Time Frame: 6 months post intervention
Population: Data were not collected from 2 participants in the attention control condition arm because they did not complete the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 22
Participants | 19 | 17

43. Secondary Outcome: Depression as Measured by Patient Health Questionnaire-9 (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) is a 9 item questionnaire. Each Item is scored from 0 (not at all) to 3 (nearly every day). The 9 items were added to generate a scale from 0 to 27, with higher scores indicating more severe depression.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 44 | 45
score on a scale | 8.23 (7.56) | 7.2 (6.47)

44. Secondary Outcome: Depression as Measured by Patient Health Questionnaire-9 (PHQ-9)
Description: as for outcome 43
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 7.5 (7.06) | 8.97 (7.14)

45. Secondary Outcome: Depression as Measured by Patient Health Questionnaire-9 (PHQ-9)
Description: as for outcome 43
Time Frame: 3 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 31 | 28
score on a scale | 6.19 (5.9) | 7.57 (8.08)

46. Secondary Outcome: Depression as Measured by Patient Health Questionnaire-9 (PHQ-9)
Description: as for outcome 43
Time Frame: 6 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 23
score on a scale | 9.52 (7.48) | 7.04 (6.2)

47. Secondary Outcome: Anxiety as Measured by Generalized Anxiety Disorder (GAD) Scale
Description: The Anxiety as Measured by Generalized Anxiety Disorder (GAD) scale is a 7 item questionnaire. Each item is scored from 0 (not at all) to 3 (nearly every day). The 7 items were added to generate a scale from 0 to 21, with higher scores indicating greater severity of symptoms of anxiety.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 44 | 45
score on a scale | 6.82 (6.06) | 5.53 (5.86)

48. Secondary Outcome: Anxiety as Measured by Generalized Anxiety Disorder (GAD) Scale
Description: as for outcome 47
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 6.81 (5.67) | 6.26 (5.96)

49. Secondary Outcome: Anxiety as Measured by Generalized Anxiety Disorder (GAD) Scale
Description: as for outcome 47
Time Frame: 3 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 31 | 28
score on a scale | 5.68 (5.53) | 5.54 (6.17)

50. Secondary Outcome: Anxiety as Measured by Generalized Anxiety Disorder (GAD) Scale
Description: as for outcome 47
Time Frame: 6 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 23
score on a scale | 8.04 (6.52) | 5.04 (4.74)

51. Secondary Outcome: Distress as Measured by PROMIS Item Bank v.1.0-Emotional Distress
Description: The Promise item bank v.1.0- Emotional Distress 7 item questionnaire includes responses from 1 (never) to 5 (always). Total score ranges from 7 to 35, a higher score indicating higher emotional distress.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 44 | 45
score on a scale | 17.55 (7.84) | 14.69 (7.77)

52. Secondary Outcome: Distress as Measured by PROMIS Item Bank v.1.0-Emotional Distress
Description: as for outcome 51
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 16.44 (7.25) | 16.4 (7.96)

53. Secondary Outcome: Distress as Measured by PROMIS Item Bank v.1.0-Emotional Distress
Description: as for outcome 51
Time Frame: 3 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 31 | 28
score on a scale | 16.19 (6.99) | 15.86 (8.63)

54. Secondary Outcome: Distress as Measured by PROMIS Item Bank v.1.0-Emotional Distress
Description: as for outcome 51
Time Frame: 6 months post intervention
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 23
score on a scale | 17.76 (7.81) | 14.39 (6.81)

55. Secondary Outcome: Risk Seeking as Measured by Risk Propensity Scale.
Description: The Risk Propensity Scale is 7 items and total score ranges from 0 to 100, a higher score indicating greater risk taking.
Time Frame: Baseline
Population: Data were not collected from 2 participants in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 43 | 45
score on a scale | 39.08 (19.08) | 40.63 (14.82)

56. Secondary Outcome: Risk Seeking as Measured by Risk Propensity Scale.
Description: as for outcome 55
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: Data were not collected from 2 participants in the tailored MBI (.b) arm because they did not complete the survey. Data were not collected from 7 participants in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 34 | 32
score on a scale | 43.32 (14.72) | 43.36 (12.95)

57. Secondary Outcome: Risk Seeking as Measured by Risk Propensity Scale.
Description: as for outcome 55
Time Frame: 3 months post intervention
Population: Data were not collected from 3 participants in the tailored MBI (.b) arm because they did not complete the survey. Data were not collected from 1 participant in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 28 | 27
score on a scale | 44.43 (14.09) | 45.56 (9.0)

58. Secondary Outcome: Risk Seeking as Measured by Risk Propensity Scale.
Description: as for outcome 55
Time Frame: 6 months post intervention
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 20
score on a scale | 40.97 (11.57) | 46.35 (8.78)

59. Secondary Outcome: Executive Function as Measured by the Amsterdam Executive Function Inventory (AEFI)
Description: Executive Function as Measured by the 13 item Amsterdam Executive Function Inventory (AEFI) total score ranges from 1 (true) to 3 (not true), higher score indicates better executive abilities.
Time Frame: Baseline
Population: Data were not collected from 1 participant in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 44 | 45
score on a scale | 2.03 (0.27) | 2.17 (0.42)

60. Secondary Outcome: Executive Function as Measured by the Amsterdam Executive Function Inventory (AEFI)
Description: as for outcome 59
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 36 | 35
score on a scale | 2.07 (0.32) | 2.05 (0.28)

61. Secondary Outcome: Executive Function as Measured by the Amsterdam Executive Function Inventory (AEFI)
Description: as for outcome 59
Time Frame: 3 months post intervention
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 30 | 27
score on a scale | 2.01 (0.28) | 2.11 (0.27)

62. Secondary Outcome: Executive Function as Measured by the Amsterdam Executive Function Inventory (AEFI)
Description: as for outcome 59
Time Frame: 6 months post intervention
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 25 | 22
score on a scale | 2.04 (0.29) | 2.05 (0.33)

63. Secondary Outcome: Positive Affect as Measured by Positive and Negative Affect Scale (PANAS-SF)
Description: PANAS-SF is a 20 item questionnaire, each item is scored from 1(very slightly or not at all)-5(extremely). Positive affect is measured by 10 items (items 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19) score ranges for 10-50 with higher scores indicating higher levels of positive effect. The Positive affect score is reported.
Time Frame: Baseline
Population: Data were not collected from 6 participants in the tailored MBI (.b) arm because they did not complete the survey. Data were not collected from 6 participants in the attention control condition arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 39 | 39
score on a scale | 31.95 (7.06) | 32.62 (12.4)

64. Secondary Outcome: Positive Affect as Measured by Positive and Negative Affect Scale (PANAS-SF)
Description: as for outcome 63
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: Data were not collected from 4 participants in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 32 | 39
score on a scale | 34.22 (9.55) | 31.49 (11.59)

65. Secondary Outcome: Negative Affect as Measured by Positive and Negative Affect Scale (PANAS-SF)
Description: PANAS-SF is a 20 item questionnaire, each item is scored from 1(very slightly or not at all)-5(extremely). Negative affect is measured by 10 items (items 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20) score ranges from 10-50, with lower scores indicating lower levels of negative effect. The negative affect score is reported.
Time Frame: Baseline
Population: as for outcome 63
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 39 | 39
score on a scale | 17.54 (7.84) | 18.1 (8.5)

66. Secondary Outcome: Negative Affect as Measured by Positive and Negative Affect Scale (PANAS-SF)
Description: as for outcome 65
Time Frame: immediately after completing the intervention (about 2 to 4 weeks after baseline)
Population: Data were not collected from 4 participants in the tailored MBI (.b) arm because they did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 32 | 39
score on a scale | 17.88 (8.21) | 18.54 (9.78)

67. Primary Outcome: Acceptability as Assessed by the Credibility and Expectancy Questionnaire - Credibility Subscale
Description: The Credibility and Expectancy Questionnaire (CEQ) was used to assess the acceptability of the intervention. All participants completed both subscales: the credibility subscale and the expectancy subscale. Each subscale total score ranges from 0 to 10, with higher scores indicating greater perceived acceptability. The credibility subscale is reported.
Time Frame: 6 months post intervention
Population: Data were only collected from participants who completed the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tailored MBI (.b) | Attention Control Condition
Number analyzed (Participants) | 32 | 29
score on a scale | 7.56 (1.53) | 6.53 (2.22)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Tailored MBI (.b) | Attention Control Condition
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT04950816/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT04950816/ICF_001.pdf